CLINICAL TRIAL: NCT03169556
Title: Comparison of Conventional Lightwand Intubation Versus Video-laryngoscope Guided Lightwand Intubation in Simulated Cervical Spine-immobilized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2016-0069
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: General Anesthesia
Keywords: Intubation; light wand; video laryngoscopy; cervical spine immobilization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video-laryngoscope guided lightwand (Experimental)
  Interventions: Device: Video-laryngoscope guided lightwand
- lightwand (Active Comparator)
  Interventions: Device: lightwand alone

INTERVENTIONS:
Device: Video-laryngoscope guided lightwand — After anesthetic induction,the difficult airway is simulated by wearing a semi-hard neck collar. For intubation, video-laryngoscope is inserted into the oral cavity ntil the epiglottis tip was visible without lifting the epiglottic vallecula. Then, the endotracheal tube with lightwand is inserted toward the midline under the epiglottis and the intubation is performed looking the transilluminated light of lightwand.
  Other Names: Video laryngoscope (VL310, Zhejiang UE Medical, Zhejiang, China)
  Arms: video-laryngoscope guided lightwand
Device: lightwand alone — After anesthetic induction,the difficult airway is simulated by wearing a semi-hard neck collar. Then, the endotracheal tube with lightwand is inserted and the intubation is performed with conventional method (blind technique by confirming transillumination).
  Other Names: LightWand (3960, GE Healthcare, Englewood, USA)
  Arms: lightwand

SUMMARY:
Among advanced intubation equipment for difficult intubation, a lighted stylet (lightwand) is a widely used equipment in cervical immobilized patients. However, a lightwand, which is used blind, is difficult to make midline positioning and can increase airway complications and hemodynamic changes. In contrast, videolaryngoscope can view vocal cord indirectly through camera, however, it requires cervical movement. Therefore, investigator hypothesized that the combined use of video-laryngoscope and lightwand for intubation can improve the efficacy of intubation compared to the use of lightwand alone in cervical immobilized patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20- 80 yrs
2. Patients scheduled surgery under the general anesthesia

Exclusion Criteria:

1. Patient who has history of gastro-esophageal reflux disease, previous airway surgery, anatomical abnormality in the upper airway, or coagulopathy
2. Patients with body mass index >35kg/m2, hemodynamic instability or loosening teeth
3. Patient who disagrees to participate this study or lacks decision-making ability, illiteracy, or foreigner
4. American Society of Anesthesiologists physical status ≥ 3

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
The success rate of intubation | Within 90 sec after insertion of lightwand or video-laryngosocpe into oral cavity.
  Confirm the success intubation through end-tidal carbon dioxide on a capnography
The duration of intubation | Within 90 sec after insertion of lightwand or video-laryngosocpe into oral cavity.
  Define as the duration between insertion of lightwand or video-laryngoscope to oral cavity and removal all intubating devices from oral cavity.

SECONDARY OUTCOMES:
number of intubation trial and scooping movements | during intubation time, intubation attempts allows maximum 3 times, within 90 sec in each time
  The number of intubation tiral and scooping movements during intubation
Blood pressure change | from start of intubation to 5minute after intubation
  The difference between maximum mean blood pressure and minimum blood pressure
Injuries of oral cavity | at immediate after intubation and extubation
  Check any blood in lips, teeth, endotracheal cuff, and oral cavity
Postoperative hoarseness | at 1hr after PACU arrival and 24hr after operation
  Check "Yes or No" through questioning the patient
Postoperative sore throat | at 1hr after PACU arrival and 24hr after operation
  Check using visual analog scale (0-100 points)
Heart rate change | from start of intubation to 5minute after intubation
  The difference between maximum heart rate and minimum minimum heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No